CLINICAL TRIAL: NCT06305000
Title: Impact of Keratinized Mucosa Augmentation Following Non-surgical Therapy on Treatment Outcomes of Peri-implant Mucositis.
Brief Title: Impact of Keratinized Mucosa Augmentation on Treatment Outcomes of Peri-implant Mucositis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Ayse Ege SELMAN, Principle Investigator, Biruni University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-KAEK-80-23-25
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Peri-implant Mucositis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Peri-implant healthy group with sufficient keratinized mucosa (≥ 2mm) (No Intervention)
- Peri-implant mucositis group with sufficient keratinized mucosa (≥ 2mm) (Experimental): Only non-surgical therapy will apply
  Interventions: Procedure: Non-surgical treatment
- Peri-implant mucositis group with insufficient keratinized mucosa (< 2mm) receiving FGG (Experimental): Free gingival graft will apply following non-surgical therapy
  Interventions: Procedure: Non-surgical treatment; Procedure: Free gingival graft

INTERVENTIONS:
Procedure: Non-surgical treatment — Non-surgical treatment consists of oral hygiene instructions, full mouth supragingival scaling using titanium hand instruments, ultrasonic devices, and subgingival debridement under local anesthesia with titanium curettes and ultrasonic instruments in a single appointment.
  Arms: Peri-implant mucositis group with insufficient keratinized mucosa (< 2mm) receiving FGG; Peri-implant mucositis group with sufficient keratinized mucosa (≥ 2mm)
Procedure: Free gingival graft — After adequate local anesthesia is achieved. A horizontal incision is placed mucogingival junction level to prepare the recipient bed. A split-thickness flap is raised without disturbing the periosteum. FGG is obtained from the palate, extending from the mesial surface of the second premolar to the middle of the first molar. The graft is shaped and stitched on the recipient surface.
  Arms: Peri-implant mucositis group with insufficient keratinized mucosa (< 2mm) receiving FGG

SUMMARY:
This study aims to observe the effects of keratinized mucosa width on peri-implant tissues by evaluating clinical and biochemical parameters. The main question it aims to answer is:

Would increasing the width of the keratinized mucosa with free gingival graft (FGG) in peri-implant mucositis be beneficial in terms of clinical periodontal parameters and peri-implant crevicular fluid levels of inflammatory cytokines compared to non-surgical therapy alone?

Our study consists of 4 groups:

Peri-implant healthy group with sufficient keratinized mucosa (≥ 2mm) (n=16), peri-implant mucositis group with sufficient keratinized mucosa (n=16), peri-implant mucositis group with insufficient keratinized mucosa (< 2mm) receiving only non-surgical treatment (n=16), peri-implant mucositis group with insufficient keratinized mucosa receiving FGG in addition to non-surgical treatment (n=16). Clinical and biochemical measurements will be recorded at the baseline, 1st month, 4th month and 7th month of the study. Peri-implant crevicular fluid samples will be collected at baseline, 1st month, 4th month and 7th month. IL-1β, RANKL, OPG levels, and RANKL/OPG ratio will be analyzed from collected samples.

Researchers will evaluate the possible benefits of FGG application in addition to non-surgical therapy by comparing the biochemical and clinical changes in areas with and without FGG application in the treatment of peri-implant mucositis.

ELIGIBILITY:
Inclusion Criteria:

* Individual dental implants with a fixed prosthetic restoration that has been functional for at least 1 year
* No systemic disease and medication use that may affect periodontal or peri-implanter tissues
* Not receiving periodontal treatment in the last 6 months
* Volunteering to participate in the study

Exclusion Criteria:

* Prosthetic restorations with an excessive contour which do not allow peri-implant pocket measurement
* Being pregnant or breastfeeding,
* Autoimmune and/or inflammatory diseases of the oral cavity,
* Active periodontal disease
* Smokers (≥ 10 cigarettes per day)
* Improperly positioned implants

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-03-27 (Actual); Primary Completion 2026-09-10 (Estimated); Study Completion 2026-09-10 (Estimated)

PRIMARY OUTCOMES:
Inflammatory parameter levels in peri-implant crevicular fluid | Baseline (prior to therapy)
  Peri-implant crevicular fluid samples will be collected from 3 sites (mesiobuccal, buccal, distobuccal) of the implants using methylcellulose strips PerioPaper® (Oralflow Inc., Smithtown, NY, USA) gently placed into the cleansed and dried pocket for 30 sec. Interleukin-1beta, RANKL and OPG levels and RANKL/ OPG ratio will be evaluated.
Inflammatory parameter levels in peri-implant crevicular fluid | 1st month
  Peri-implant crevicular fluid samples will be collected from 3 sites (mesiobuccal, buccal, distobuccal) of the implants using methylcellulose strips PerioPaper® (Oralflow Inc., Smithtown, NY, USA) gently placed into the cleansed and dried pocket for 30 sec. Interleukin-1beta, RANKL and OPG levels and RANKL/ OPG ratio will be evaluated.
Inflammatory parameter levels in peri-implant crevicular fluid | 4th month
  Peri-implant crevicular fluid samples will be collected from 3 sites (mesiobuccal, buccal, distobuccal) of the implants using methylcellulose strips PerioPaper® (Oralflow Inc., Smithtown, NY, USA) gently placed into the cleansed and dried pocket for 30 sec. Interleukin-1beta, RANKL and OPG levels and RANKL/ OPG ratio will be evaluated.
Inflammatory parameter levels in peri-implant crevicular fluid | 7th month
  Peri-implant crevicular fluid samples will be collected from 3 sites (mesiobuccal, buccal, distobuccal) of the implants using methylcellulose strips PerioPaper® (Oralflow Inc., Smithtown, NY, USA) gently placed into the cleansed and dried pocket for 30 sec. Interleukin-1beta, RANKL and OPG levels and RANKL/ OPG ratio will be evaluated.

SECONDARY OUTCOMES:
Plaque index (Silness & Löe, 1964) | Baseline (prior to therapy)
  0: Absence of microbial plaque
  1. Thin plaque layer at the mucosal margin, only detectable by scraping with a probe
  2. Moderate layer of plaque in the along the mucosal margin; interdental spaces free, but plaque is visible to naked eye
  3. Abundant plaque along with the mucosal margin; interdental places filled with plaque
Plaque index (Silness & Löe, 1964) | 1st month
  Plaque index (Silness & Löe, 1964):
  0: Absence of microbial plaque
  1. Thin plaque layer at the mucosal margin, only detectable by scraping with a probe
  2. Moderate layer of plaque in the along the mucosal margin; interdental spaces free, but plaque is visible to naked eye
  3. Abundant plaque along with the mucosal margin; interdental places filled with plaque
Plaque index (Silness & Löe, 1964) | 4th month
  0: Absence of microbial plaque
  1. Thin plaque layer at the mucosal margin, only detectable by scraping with a probe
  2. Moderate layer of plaque in the along the mucosal margin; interdental spaces free, but plaque is visible to naked eye
  3. Abundant plaque along with the mucosal margin; interdental places filled with plaque
Plaque index (Silness & Löe, 1964) | 7th month
  0: Absence of microbial plaque
  1. Thin plaque layer at the mucosal margin, only detectable by scraping with a probe
  2. Moderate layer of plaque in the along the mucosal margin; interdental spaces free, but plaque is visible to naked eye
  3. Abundant plaque along with the mucosal margin; interdental places filled with plaque
Gingival Index ( Löe & Silness,1963) | Baseline (prior to therapy)
  0: normal gingiva
  1. mild inflammation - slight change in color and slight edema but no bleeding on probing
  2. moderate inflammation - redness, edema and glazing, bleeding on probing
  3. severe inflammation - marked redness and edema, ulceration with tendency to spontaneous bleeding
Gingival Index ( Löe & Silness,1963) | 1st month
  0: normal gingiva
  1. mild inflammation - slight change in color and slight edema but no bleeding on probing
  2. moderate inflammation - redness, edema and glazing, bleeding on probing
  3. severe inflammation - marked redness and edema, ulceration with tendency to spontaneous bleeding
Gingival Index ( Löe & Silness,1963) | 4th month
  0: normal gingiva
  1. mild inflammation - slight change in color and slight edema but no bleeding on probing
  2. moderate inflammation - redness, edema and glazing, bleeding on probing
  3. severe inflammation - marked redness and edema, ulceration with tendency to spontaneous bleeding
Gingival Index ( Löe & Silness,1963) | 7th month
  0: normal gingiva
  1. mild inflammation - slight change in color and slight edema but no bleeding on probing
  2. moderate inflammation - redness, edema and glazing, bleeding on probing
  3. severe inflammation - marked redness and edema, ulceration with tendency to spontaneous bleeding
Bleeding on probing (Ainamo & Bay 1975) | Baseline (prior to therapy)
  Bleeding on probing A bleeding-on-probing percentage score assessed as the proportion of bleeding sites (dichotomous yes/no evaluation) when stimulated by a standardized manual probe with a controlled (~25 g) force to the bottom of the sulcus/pocket at six sites (mesiobuccal, buccal, distobuccal, mesiolingual, lingual, distolingual) on all present teeth/ implants.
Bleeding on probing (Ainamo & Bay 1975) | 1st month
  Bleeding on probing A bleeding-on-probing percentage score assessed as the proportion of bleeding sites (dichotomous yes/no evaluation) when stimulated by a standardized manual probe with a controlled (~25 g) force to the bottom of the sulcus/pocket at six sites (mesiobuccal, buccal, distobuccal, mesiolingual, lingual, distolingual) on all present teeth/ implants.
Bleeding on probing (Ainamo & Bay 1975) | 4th month
  Bleeding on probing A bleeding-on-probing percentage score assessed as the proportion of bleeding sites (dichotomous yes/no evaluation) when stimulated by a standardized manual probe with a controlled (~25 g) force to the bottom of the sulcus/pocket at six sites (mesiobuccal, buccal, distobuccal, mesiolingual, lingual, distolingual) on all present teeth/ implants.
Bleeding on probing (Ainamo & Bay 1975) | 7th month
  Bleeding on probing A bleeding-on-probing percentage score assessed as the proportion of bleeding sites (dichotomous yes/no evaluation) when stimulated by a standardized manual probe with a controlled (~25 g) force to the bottom of the sulcus/pocket at six sites (mesiobuccal, buccal, distobuccal, mesiolingual, lingual, distolingual) on all present teeth/ implants.
Keratinized mucosa width | Baseline (prior to therapy)
  The apical-coronal distance from the mucosal margin to the mucogingival junction (MGJ) Measurements will be made at three points on implants (mesiobuccal, midbuccal, distobuccal) using a periodontal probe.
Keratinized mucosa width | 1st month
  The apical-coronal distance from the mucosal margin to the mucogingival junction (MGJ). Measurements will be made at three points on implants (mesiobuccal, midbuccal, distobuccal) using a periodontal probe.
Keratinized mucosa width | 4th month
  The apical-coronal distance from the mucosal margin to the mucogingival junction (MGJ). Measurements will be made at three points on implants (mesiobuccal, midbuccal, distobuccal) using a periodontal probe.
Keratinized mucosa width | 7th month
  The apical-coronal distance from the mucosal margin to the mucogingival junction (MGJ). Measurements will be made at three points on implants (mesiobuccal, midbuccal, distobuccal) using a periodontal probe.
Probing depth | Baseline (prior to therapy)
  Probing pocket depth: The distance from the base of the pocket to the mucosal margin. Measurements will be made at six points on all teeth/ implants (mesiobuccal, midbuccal, distobuccal, mesiolingual, midlingual, and distolingual) using a periodontal probe.
Probing depth | 1st month
  Probing pocket depth: The distance from the base of the pocket to the mucosal margin. Measurements will be made at six points on all teeth/ implants (mesiobuccal, midbuccal, distobuccal, mesiolingual, midlingual, and distolingual) using a periodontal probe.
Probing depth | 4th month
  The distance from the base of the pocket to the mucosal margin. Measurements will be made at six points on all teeth/ implants (mesiobuccal, midbuccal, distobuccal, mesiolingual, midlingual, and distolingual) using a periodontal probe.
Probing depth | 7th month
  The distance from the base of the pocket to the mucosal margin. Measurements will be made at six points on all teeth/ implants (mesiobuccal, midbuccal, distobuccal, mesiolingual, midlingual, and distolingual) using a periodontal probe.

CONTACTS AND LOCATIONS:
Overall Officials: Ayse E Selman, Principal Investigator — Biruni University
Locations (1):
- Biruni University, Istanbul, Turkey (Türkiye)